CLINICAL TRIAL: NCT06130748
Title: Effectiveness of Two Mini-screws Supported Hyrax for Maxillary Expansion in Early Adulthood: A Randomized Control Trial.
Brief Title: Effectiveness of Two Mini-screws Supported Hyrax for Maxillary Expansion in Early Adulthood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, abdullah mohammed ali al-thalabi, Master Degree student ,Faculty of Dentistry ,Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15623
Record Dates: First submitted 2023-11-03; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Transverse Maxillary Deficiency
Keywords: maxillary expansion

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Hyrax (Experimental): Device: Hybrid hyrax these patents will be treated using Two mini-screws supported hybrid hyrax
  Other Names:
  • MARPE(miniscrews-assisted rapid palatal expander)
  Interventions: Device: Hybrid Hyrax
- Untreated control group (No Intervention): Ethically ,these patents will be treated at the end of the study using the same appliance used for the experimental group

INTERVENTIONS:
Device: Hybrid Hyrax — these patents will be treated using Two mini-screws supported hybrid hyrax
  Other Names: MARPE(miniscrews-assisted rapid palatal expander)
  Arms: Hybrid Hyrax

SUMMARY:
The study aiming at evaluation of the Skeletal and Dento-alveolar expansion in adult patents using Two Mini-screws Supported Hyrax compared with untreated control group.

DETAILED DESCRIPTION:
Methodology:

* Basic orthodontic record will be taken.
* impression with bands on upper first molars will be taken.
* Two eyelets will be soldered to the body of the hyrax appliance (size 10, Dentaurum, Germany).
* CBCT will be taken while patient wearing 1 mm thickness vacuum on the lower arch to dis-occlude both arches.
* Delivery, check the retention and fitness of the appliance.
* Cementation of the appliance using band cement(compomer).
* Using 3M contra-angle driver, the screws (Tomas screw size 10, Dentaurum, Germany) will be loaded and inserted.
* Activation of the appliance by opening it two turns immediately, followed by two turns everyday till cross bite correction or appearance of midline diastema.
* Closure of the device, and leave the appliance in-situ for five months as a retention.
* Post-expansion CBCT will be taken and continue fixed orthodontic treatment. Outcome: skeletal and dento-alveolar expansion will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral Dental posterior cross-bite
* Skeletal Maxillary constriction
* Male and female patients.
* Chronological age (18-30 years).
* Mid-palatal suture maturation (Grade C,D ) according to F Angileri classification
* Good oral hygiene.
* No craniofacial anomalies or syndromes

Exclusion Criteria:

* Scissor-bite
* Orthodontically-treated
* functional cross bite due to premature occlusal contact
* patients with a syndrome
* cleft patients

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Skeletal maxillary expansion To compare the amount of skeletal expansion pre and post expansion | the outcome will be assessed five months post-expansion
  To compare the amount of skeletal expansion using linear and angular measurements and the expansion pattern of mid-palatal suture extracted from cone beam computed tomography pre and post expansion

SECONDARY OUTCOMES:
Dento-alaveolar expansion | the outcome will be assessed five months post-expansion
  To compare the amount of dento-alveolar expansion using linear and angular measurements extracted from cone beam computed tomography pre and post-expansion

CONTACTS AND LOCATIONS:
Overall Officials: abdullah mo ali al-thalabi, Msc candidate, Principal Investigator — Cairo University
Locations (1):
- faculty of dentistry, Cairo university, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided